CLINICAL TRIAL: NCT04673240
Title: CLINICAL EFFECT OF BOTULINUM TOXIN TYPE A IN THE TREATMENT OF SPASTICITY AFTER TRAUMATIC BRAIN INJURY, SPINAL CORD INJURY OR IN MULTIPLE SCLEROSIS PATIENTS: AN OBSERVATIONAL STUDY
Brief Title: CLINICAL EFFECT OF BOTULINUM TOXIN TYPE A IN TREATMENT OF SPASTICITY
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other)
Collaborators: Ipsen (Industry); Azienda Ospedaliero Universitaria Maggiore della Carita (Other); SIRN (Unknown)
Responsible Party: Principal Investigator, Alessio Baricich, MD PhD, Università degli Studi del Piemonte Orientale Amedeo Avogadro
Other Study IDs: NSS_BoNT-A
Record Dates: First submitted 2020-12-12; First posted 2020-12-17 (Actual); Last update posted 2020-12-17 (Actual); Status verified 2020-12

CONDITIONS: Spasticity; Brain Injuries; Spinal Cord Injuries; Multiple Sclerosis
MeSH Terms: conditions — Muscle Spasticity; Brain Injuries; Spinal Cord Injuries; Multiple Sclerosis | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: US Export: No

INTERVENTIONS:
Drug: Botulinum toxin type A injection — Adult patients with spasticity due to traumatic brain injury, spinal cord injury, or MS, treated with Botulinum Toxin type A.
  As this is a non-interventional study, no diagnostic, therapeutic, or experimental intervention is involved. Subjects will receive clinical assessments, medications, and treatments solely as determined by their study physician.

SUMMARY:
Spasticity has been defined as a disorder of the sensorimotor system characterized by a velocity-dependent increase in tonic stretch reflexes (muscle tone) with exaggerated tendon jerks, resulting from hyperexcitability of the stretch reflex.

The treatment goal of spasticity is Medical treatment generally combines physiotherapy with medications, depending on spasticity distribution. Systemic treatments such as oral or intrathecal baclofen are generally considered in case of generalized spasticity, whereas local treatments are considered in case of focal spasticity.

Local treatments such as Botulinum Toxin type A, phenol, and alcohol present several advantages, allowing to treat of selected muscles without the risk of sedation. As stated above, they are indicated for focal spasticity but might be helpful even in the presence of generalized spasticity with identified focal goals (Bethoux et al., 2015).

In particular, Botulinum Toxin type A (BoNT-A) is considered the gold standard treatment for focal spasticity, showing a level A evidence for spasticity reduction in upper- and lower-limb spasticity (Simpson et al., 2016).

However, current evidence is mainly focused on post-stroke spasticity (Franceschini et al., 2014), whereas it is still limited in spasticity as a consequence of other aetiologies, such as spinal cord injury (SCI), traumatic brain injury (TBI), or multiple sclerosis (MS).

Interestingly, spasticity is a major concern for the rehabilitation of these patients.

The aim of this observational study is the evaluation of the clinical efficacy of BoNT-A in spasticity reduction in patients affected by neurological conditions different from post-stroke spasticity, such as SCI, TBI, and MS.

ELIGIBILITY:
Inclusion Criteria:

* Age >18 years
* Spasticity as a consequence of traumatic brain injury, spinal cord injury or MS (documented by clinical records)
* Muscle tone graded at least 1+ on the modified Ashworth scale in the relevant joints of the affected limb(s), which requires medical intervention
* BoNT naïve or pre-treated with any BoNT product. If previously treated with any BoNT, at least a 4 months interval between last injection and inclusion

Exclusion Criteria:

* Presence of fixed contractures or bony deformities in the affected limb
* Changes in any oral antispastic medications or specific physiotherapy regimen <4m before study entry or during the study.
* Other neurological or orthopaedic conditions involving the affected limbs.
* Sensitivity to BoNT-A or to its excipients
* Other contraindications as given in the local SmPC for BoNT-A

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients with spasticity as a consequence of traumatic brain injury, spinal cord injury or MS, treated with Botulinum Toxin type A.
Sampling Method: Probability Sample
Enrollment: 70 (Estimated)
Dates: Start 2019-03-29 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2022-06-30 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale (MAS) | 1 month
  Percentage of patients with at least 1 point reduction of MAS in any treated muscle, 1 month after BoNT-A injection injection of Botulinum toxin A (responders)

SECONDARY OUTCOMES:
Global Assessment of Efficacy scale) | 1 month and 3 months after boNT-A injection
  Evaluation of treatment goal achievement by the physicians, patients and caregivers at 1 and 3 months after BoNT-A injection
active range of motion | e, 1, 3 and 6 months or before new BoNT-A injection
  Documentation of active range of motion (a-ROM) for the treated joints in the overall study population at baseline, 1, 3 and 6 months or before new BoNT-A injection using a handheld goniometer.
passive range of motion | e, 1, 3 and 6 months or before new BoNT-A injection
  Documentation of passive range of motion (p-ROM) for the treated joints in the overall study population at baseline, 1, 3 and 6 months or before new BoNT-A injection using a handheld goniometer.
Numeric Rating Scale for pain | , 1, 3 and 6 months after BoNT-A or before the new BoNT-A injection
  Pain will be assessed in the overall study population at baseline, 1, 3 and 6 months after BoNT-A or before the new BoNT-A injection using Numeric Rating Scale (pain).
EQ5-D | 1, 3 and 6 months after BoNT-A or before the new BoNT-A injection
  Quality of life will be assessed in the overall study population at baseline, 1, 3 and 6 months after BoNT-A or before the new BoNT-A injection using EQ5-D questionnaire.
interval of time between BoNT-A reinjections | 3-6 months
  Documentation of the interval of time between reinjections will be assessed during 6-months follow up (if applicable)

CONTACTS AND LOCATIONS:
Overall Officials: Alessio Baricich, Study Chair — Università del Piemonte orientale "Amedeo Avogadro"
Locations (1):
- Azienda Ospedaliero Universitaria Maggiore della Carità, Novara, Italy

REFERENCES:
- [Derived] Baricich A, Battaglia M, Cuneo D, Cosenza L, Millevolte M, Cosma M, Filippetti M, Dalise S, Azzollini V, Chisari C, Spina S, Cinone N, Scotti L, Invernizzi M, Paolucci S, Picelli A, Santamato A. Clinical efficacy of botulinum toxin type A in patients with traumatic brain injury, spinal cord injury, or multiple sclerosis: An observational longitudinal study. Front Neurol. 2023 Apr 6;14:1133390. doi: 10.3389/fneur.2023.1133390. eCollection 2023. PMID 37090974